CLINICAL TRIAL: NCT04690166
Title: Validation and Cultural Adaptation of the Turkish Translation of the London Speech Evaluation Scale
Brief Title: Validation of the Turkish Translation of the London Speech Evaluation Scale
Status: Completed | Type: Observational
Sponsor: Prof. Dr. Cemil Tascıoglu Education and Research Hospital Organization (Other)
Responsible Party: Principal Investigator, Yavuz Atar, Associate Professor, M.D., Prof. Dr. Cemil Tascıoglu Education and Research Hospital Organization
Other Study IDs: 462
Record Dates: First submitted 2020-12-26; First posted 2020-12-30 (Actual); Last update posted 2021-07-29 (Actual); Status verified 2021-07

CONDITIONS: Speech Intelligibility; Speech Disorders; Head and Neck Cancer; Speech Dysfunction; Speech
Keywords: Perceptual; speech; articulation; neck; cancer
MeSH Terms: conditions — Speech Intelligibility; Speech Disorders; Head and Neck Neoplasms; Speech; Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cancer Patients: In outpatients clinic, the first group consists of 60 head and neck cancer patients who were treated by ours. The participants will given the document consists that "bit, bet, but" words and also a brief part of "Diyet passage" who written by Omer Seyffettin. The speech record of patients who read to document, will evaluated by three judges (otorhinolaryngologist). Three judges will scoring to Turkish translation of London Speech Evaluation Scale (LSE-T), consists of 6 parameters. After the six weeks, the records were scored again as randomisely.
  Interventions: Other: The speech records related to the reading document
- Healty Control: In outpatients clinic, the control group consists of 60 patients who have not speech and hear impairments. The participants will given the document consists that "bit, bet, but" words and also a brief part of "Diyet passage" who written by Omer Seyffettin. The speech record of patients who read to document, will evaluated by three judges (otorhinolaryngologist). Three judges will scoring to Turkish translation of London Speech Evaluation Scale (LSE-T), consists of 6 parameters. After the six weeks, the records were scored again as randomisely.
  Interventions: Other: The speech records related to the reading document

INTERVENTIONS:
Other: The speech records related to the reading document — The document consists "bit, bet, but" words and Diyet passage. Volunteers will read the document in front of the microphone and also the speech will recorded by a computer.

SUMMARY:
Purpose of the study is the validation and cultual adaptation of the Turkish translation of the London Speech Evaluation Scale (LSE-T), so that it would be used as an assessment tool for Turkish head and neck cancer patients. There is no validated Turkish version of LSE to measure severity of perceptual speech in head and neck cancer patients.

DETAILED DESCRIPTION:
The speech function is a multidirectional process that depends on complex neuro-muscular network. The function can be evaluated using instrumental, such as voice analysis computer programmes, scales, or well structured questionnaires. There are many scales for assessment of perceptual speech but there is no validated for head and neck patients. The study will assess the construct validity and adaptation of the Turkish translation of Speech Specific Perceptual Speech Evaluation as known as London Speech Evaluation Scale. The investigators developed the Turkish translation of this scale (LSE-T), according to the cross-cultural adaptation guidelines. Two translators translated the LSE into Turkish and a native English language speaker reverse-translated it into English. The back translation was sent to the original author for proofreading. The LSE scale consisted of 6 parameters and 4 scores related with perceptual speech in head and neck cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Able to speak, read, understand and write in Turkish
* History of oral, orofarengeal cancer
* Volunteers who accept the informed consent

Exclusion Criteria:

* Mental disorders
* Cognitive limitations
* Able not to speak, read, understand and write in Turkish
* Underwent any surgery last six month
* Permanent tracheostomy, total laryngectomy
* Pregnancy
* Out of age 18-70 years old
* Adults who do not accept the informed consent.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults with oral, oropharyngeal cancer and healthy adults
Sampling Method: Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2020-12-21 (Actual); Primary Completion 2021-05-21 (Actual); Study Completion 2021-05-21 (Actual)

PRIMARY OUTCOMES:
Validation of the Turkish Translation of London Speech Evaluation Scale | Baseline
  Turkish Translation of London Speech Evaluation Scale consists of 6 parameters and 4 scores. The minimum score is 0 and maximum score is 24. The lower scores mean a better than high scores.
Validation of the Turkish Translation of London Speech Evaluation Scale | 6 weeks
  Turkish Translation of London Speech Evaluation Scale consists of 6 parameters and 4 scores. The minimum score is 0 and maximum score is 24. The lower scores mean a better than high scores.

CONTACTS AND LOCATIONS:
Overall Officials: Ziya Salturk, Asso Prof,MD, Principal Investigator — Anadolu Medical Center, In Affiliation with Johns Hopkins Medicine
Locations (1):
- Prof Dr Cemil Tascioglu City Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dwivedi RC, Rose SS, Chisholm EJ, Kerawala CJ, Clarke PM, Nutting CM, Rhys-Evans PH, Harrington KJ, Kazi R. Development and validation of first-ever speech-specific perceptual speech evaluation tool for patients with head and neck cancer: the London speech evaluation (LSE) scale. Head Neck. 2012 Jan;34(1):94-103. doi: 10.1002/hed.21683. Epub 2011 Apr 5. PMID 21469245